CLINICAL TRIAL: NCT04727749
Title: A Study of the Pawsitive Impacts of Therapy Dog Visits With Adult Emergency Department Pain Patients
Brief Title: Pawsitive Impacts of Therapy Dog Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation (Other)
Responsible Party: Principal Investigator, Colleen Dell, Research Chair in One Health & Wellness, Professor, Tenured, University of Saskatchewan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1253
Record Dates: First submitted 2021-01-22; First posted 2021-01-27 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Pain; Pain, Acute; Pain, Chronic; Pain, Intractable
Keywords: Pain; Emergency Department; Therapy Dog
MeSH Terms: conditions — Pain; Acute Pain; Chronic Pain; Pain, Intractable; Emergencies

STUDY DESIGN:
Intervention Model Description: Data is to be collected 5 days a week, with animal testing days alternating with control days.
Who Masked: Participant
Masking Description: Consent will be obtained using a deceptive consent form, which will explain that this is a pain study, but will omit any information regarding therapy dogs. Once all measures are taken, the participants will be explained the deception and asked to sign the true consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapy Dog Team Visit (Experimental): Patient interacts with the therapy dog and handler.
  Interventions: Behavioral: Therapy Dog Team Visit
- No Therapy Dog Team Visit (No Intervention): No patient interaction with the therapy dog or handler.

INTERVENTIONS:
Behavioral: Therapy Dog Team Visit — For the intervention group, patient interacts with the therapy dog, handler shares information about the therapy dog, asks about patient's pets, and offers a trading card of the therapy dog at the conclusion of the visit.
  Arms: Therapy Dog Team Visit

SUMMARY:
The goal of this unique 18 month study is to better understand the experiences of pain patients in the Royal University Hospital (RUH) Emergency Department (ED), to create excellence in health care. The purpose is to measure the impact of visiting therapy dogs on reducing ED patient pain.

DETAILED DESCRIPTION:
The goal of this unique 18 month study is to better understand the experiences of pain patients in the Royal University Hospital (RUH) Emergency Department (ED), to create excellence in health care. The purpose is to measure the impact of visiting therapy dogs on reducing ED patient pain.

The background rationale is that pain is the primary reason individuals attend an ED, patient pain is generally not well managed in EDs, Saskatchewan EDs have among the longest wait times in the country, and anxiety associated with ED waiting can negatively impact patients' pain.

Research suggests a therapy dog can change patients' perceptions of pain and its intensity and facilitate relaxation. The intervention will be examined for its impact on patients' sensory pain (i.e., physical pain severity), affective pain (i.e., emotional pain unpleasantness) and anxiety.

It is important to find creative, low-cost ways to respond to patients attending the ED for pain. The primary objective of this study is to generate new health-related knowledge on the ED pain patient experience. The secondary objectives are to implement effective end-of-grant knowledge translation and dissemination strategies and undertake a successful model of collaborative, multidisciplinary research among researchers, patient advisors and system representatives, rooted in a One Health framework.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Able to provide consent
* Attending the Emergency Department because of pain/discomfort
* Canadian Triage and Acuity Score (CTAS) of 2-5
* Willing to visit with a therapy dog team (intervention group only)

Exclusion Criteria:

* Pain medications (specifically immediate release acetaminophen and opioid analgesics) within an hour prior to the visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Dell, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carey B, Dell CA, Stempien J, Tupper S, Rohr B, Carr E, Cruz M, Acoose S, Butt P, Broberg L, Collard L, Fele-Slaferek L, Fornssler C, Goodridge D, Gunderson J, McKenzie H, Rubin J, Shand J, Smith J, Trask J, Ukrainetz K, Meier S. Outcomes of a controlled trial with visiting therapy dog teams on pain in adults in an emergency department. PLoS One. 2022 Mar 9;17(3):e0262599. doi: 10.1371/journal.pone.0262599. eCollection 2022. PMID 35263346

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at the Emergency Department of the Royal University Hospital in Saskatoon, SK, between June and September of 2019.
Period: Overall Study
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
Started | 107 | 104
Completed | 97 | 101
Not Completed | 10 | 3
Not completed — Lost to Follow-up | 10 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit | Total
Number analyzed (Participants) | 107 | 104 | 211
Age, Continuous [Median (Full Range); unit: years] | 60 [18 to 96] | 63 [18 to 95] | 62 [18 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 47 | 94
  Male | 60 | 57 | 117
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnic Origin: Aboriginal Peoples of North America | 9 | 16 | 25
  Ethnic Origin: Black | 2 | 1 | 3
  Ethnic Origin: Filipino | 1 | 3 | 4
  Ethnic Origin: South Asian | 0 | 1 | 1
  Ethnic Origin: White | 95 | 81 | 176
  Ethnic Origin: White, Aboriginal Peoples of North America | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 109 | 102 | 211
Pain Score (ESAS-r) A higher number represents a worse outcome [Count of Participants; unit: Participants]
  0 | 43 | 43 | 86
  1 | 6 | 7 | 13
  2 | 9 | 11 | 20
  3 | 7 | 8 | 15
  4 | 4 | 9 | 13
  5 | 7 | 8 | 15
  6 | 11 | 5 | 16
  7 | 5 | 6 | 11
  8 | 6 | 3 | 9
  9 | 3 | 3 | 6
  10 | 6 | 1 | 7
Anxiety Score (ESAS-r) A higher number represents a worse outcome [Count of Participants; unit: Participants]
  0 | 36 | 43 | 79
  1 | 9 | 11 | 20
  2 | 7 | 12 | 19
  3 | 6 | 9 | 15
  4 | 11 | 2 | 13
  5 | 9 | 11 | 20
  6 | 11 | 4 | 15
  7 | 7 | 3 | 10
  8 | 7 | 2 | 9
  9 | 0 | 0 | 0
  10 | 4 | 7 | 11
Depression Score (ESAS-r) A higher number represents a worse outcome [Count of Participants; unit: Participants]
  0 | 52 | 59 | 111
  1 | 4 | 6 | 10
  2 | 9 | 8 | 17
  3 | 13 | 3 | 16
  4 | 5 | 2 | 7
  5 | 3 | 9 | 12
  6 | 7 | 4 | 11
  7 | 2 | 2 | 4
  8 | 6 | 4 | 10
  9 | 1 | 5 | 6
  10 | 5 | 2 | 7
Well-being Score (ESAS-r) A higher number represents a worse outcome [Count of Participants; unit: Participants]
  0 | 6 | 13 | 19
  1 | 5 | 6 | 11
  2 | 7 | 16 | 23
  3 | 18 | 8 | 26
  4 | 11 | 12 | 23
  5 | 17 | 25 | 42
  6 | 13 | 7 | 20
  7 | 16 | 8 | 24
  8 | 6 | 3 | 9
  9 | 2 | 3 | 5
  10 | 5 | 3 | 8
Blood Pressure [Median (Full Range); unit: mm HG]
  Systolic | 126 [80 to 189] | 129 [89 to 174] | 127 [80 to 189]
  Diastolic | 74 [45 to 104] | 73 [39 to 132] | 73 [39 to 132]
Heart Rate [Median (Full Range); unit: bpm] | 77 [48 to 141] | 77 [41 to 163] | 77 [41 to 163]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Stratified by Edmonton Symptom Assessment System (Revised Version) (ESAS-r) Pain Scores
Description: Participants Stratified by Pain scores Edmonton Symptom Assessment System (revised version) (ESAS-r) 11-point rating scale (scale of 0 to 10), in which higher ratings indicate worse outcomes, Pain Scores at 20 Minutes Post Visit.
Time Frame: 20 minutes post visit
Measure: Count of Participants; unit: Participants
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
Number analyzed (Participants) | 97 | 101
Participants
  0 | 50 | 43
  1 | 7 | 7
  2 | 3 | 13
  3 | 5 | 3
  4 | 7 | 11
  5 | 7 | 7
  6 | 4 | 4
  7 | 9 | 4
  8 | 4 | 3
  9 | 0 | 6
  10 | 1 | 0

2. Primary Outcome: Change in Pain Score
Description: Pain score using the Edmonton Symptom Assessment System (revised version) (ESAS-r) 11-point rating scale (scale of 0 to 10), in which higher ratings indicate worse outcomes.
Time Frame: Baseline visit compared to 20 minutes post-visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
Number analyzed (Participants) | 97 | 101
units on a scale | -0.90 (2.05) | 0.03 (2.30)

3. Secondary Outcome: Number of Participants Stratified by Edmonton Symptom Assessment System (Revised Version) (ESAS-r) Anxiety Scores
Description: Participants Stratified by Edmonton Symptom Assessment System (revised version) (ESAS-r) 11-point rating scale (scale of 0 to 10), in which higher ratings indicate worse outcomes, Anxiety Scores at 20 Minutes Post Visit
Time Frame: 20 minutes post-visit
Measure: Count of Participants; unit: Participants
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
Number analyzed (Participants) | 97 | 101
Participants
  0 | 55 | 45
  1 | 3 | 7
  2 | 6 | 13
  3 | 11 | 8
  4 | 4 | 6
  5 | 8 | 9
  6 | 1 | 3
  7 | 5 | 2
  8 | 3 | 4
  9 | 0 | 0
  10 | 1 | 5

4. Secondary Outcome: Number of Participants Stratified by Edmonton Symptom Assessment System (Revised Version) (ESAS-r) Depression Scores
Description: Participants Stratified by Edmonton Symptom Assessment System (revised version) (ESAS-r) 11-point rating scale (scale of 0 to 10), in which higher ratings indicate worse outcomes, Depression Scores at 20 Minutes Post Visit
Time Frame: 20 minutes post-visit
Measure: Count of Participants; unit: Participants
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
Number analyzed (Participants) | 97 | 101
Participants
  0 | 51 | 55
  1 | 5 | 7
  2 | 5 | 7
  3 | 7 | 7
  4 | 7 | 5
  5 | 4 | 5
  6 | 6 | 1
  7 | 0 | 2
  8 | 4 | 6
  9 | 0 | 3
  10 | 1 | 2

5. Secondary Outcome: Number of Participants Stratified by Edmonton Symptom Assessment System (Revised Version) (ESAS-r) Well-Being Scores
Description: Participants Stratified by Edmonton Symptom Assessment System (revised version) (ESAS-r) 11-point rating scale (scale of 0 to 10), in which higher ratings indicate worse outcomes, Well-being Scores at 20 Minutes Post Visit.
Time Frame: 20 minutes post-visit
Measure: Count of Participants; unit: Participants
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
Number analyzed (Participants) | 97 | 101
Participants
  0 | 14 | 15
  1 | 5 | 6
  2 | 8 | 8
  3 | 12 | 12
  4 | 12 | 11
  5 | 26 | 26
  6 | 6 | 7
  7 | 7 | 7
  8 | 5 | 5
  9 | 2 | 2
  10 | 0 | 0

6. Secondary Outcome: Change in Blood Pressure
Description: Mean arterial blood pressure using a blood pressure cuff
Time Frame: 20 minutes post-visit
Measure: Mean (Standard Deviation); unit: mm HG
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
Number analyzed (Participants) | 97 | 101
mm HG | 1.01 (10.7) | -.04 (8.07)

7. Secondary Outcome: Change in Heart Rate
Description: Radial pulse
Time Frame: 20 minutes post-visit
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
Number analyzed (Participants) | 97 | 101
BPM | .48 (11.68) | -.4 (8.02)

8. Post Hoc Outcome: Change in Anxiety Score
Description: Anxiety score is measured using the Edmonton Symptom Assessment System (revised version) (ESAS-r) 11-point rating scale (scale of 0 to 10), in which higher ratings indicate worse outcomes.
Time Frame: Baseline visit compared to 20 minutes post-visit
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Therapy Dog Team Visit: Patient interacts with the therapy dog and handler. Therapy Dog Team Visit: For the intervention group, the patient interacts with the therapy dog, the handler shares information about the therapy dog, asks about the patient's pets, and offers a trading card of the therapy dog at the conclusion of the visit.
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
Number analyzed (Participants) | 97 | 101
units on a scale | -1.13 (2.46) | -0.11 (2.60)

9. Post Hoc Outcome: Change in Depression Score
Description: Depression score using the Edmonton Symptom Assessment System (revised version) (ESAS-r) 11-point rating scale (scale of 0 to 10), in which higher ratings indicate worse outcomes.
Time Frame: Baseline visit compared to 20 minutes post-visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
Number analyzed (Participants) | 97 | 101
units on a scale | -0.72 (1.71) | 0.02 (1.77)

10. Post Hoc Outcome: Change in Well-Being Score
Description: Well-Being score using the Edmonton Symptom Assessment System (revised version) (ESAS-r) 11-point rating scale (scale of 0 to 10), in which higher ratings indicate worse outcomes.
Time Frame: Baseline visit compared to 20 minutes post-visit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
Number analyzed (Participants) | 97 | 101
units on a scale | -0.87 (1.84) | 0.14 (1.84)

ADVERSE EVENTS:
Description: Death, serious adverse effects, and other (non-serious adverse effects) were not assessed for this study. An intervention of interaction with a therapy dog is not expected to put participants at risk of Serious Adverse Events, All-Cause Mortality, or Other.
Arm/Group | Therapy Dog Team Visit | No Therapy Dog Team Visit
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
1. Did not account for impact of handlers in therapy dog visits
2. Power analysis and larger sample needed to examine interaction of key demographic independent variables - dog experience and intersecting identity factors (ethnicity and age)
3. Intervention group of human visitation without dog not included
4. Limited to one hospital setting
5. Did not ask about medications taken at home that may have influenced pain scores
6. Various variables can influence blood pressure and heart rate

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-04-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT04727749/Prot_000.pdf